CLINICAL TRIAL: NCT03078361
Title: Latinos CARES (Colorectal Cancer Awareness, Research, Education and Screening) Project
Brief Title: Latinos CARES (Colorectal Cancer Awareness, Research, Education and Screening)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Florida Department of Health (Other Government); Bankhead-Coley Cancer Research Program (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: MCC-17665
Record Dates: First submitted 2017-03-03; First posted 2017-03-13 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2022-08

CONDITIONS: Colorectal Cancer; Colorectal Carcinoma
Keywords: cancer screening; colon
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Receptor Protein-Tyrosine Kinases

STUDY DESIGN:
Intervention Model Description: After completion of baseline assessments, participants will be randomized so that the study personnel are unaware of the intervention assignment at the time of the baseline assessment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LATINOS CARES Toolkit (Active Comparator): Participants assigned to the LATINOS CARES condition will receive an I-FOBT kit, DVD and photonovella booklet from the study coordinator. The participant will view the DVD in a private area (headphones are available) using a portable DVD player in clinic before seeing the provider. The DVD will be about 8-10 minutes long. The participant will take the LATINOS CARES toolkit and I-FOBT home after the clinic visit. The participant will be instructed to re-review the materials and complete the I-FOBT stool sampling at home.
  Interventions: Other: Immunochemical Fecal Occult Blood Test (I-FOBT) Kit; Behavioral: LATINOS CARES Toolkit
- Standard Intervention (SI) (Active Comparator): Participants assigned to the standard brochure (SI) will be provided a packet containing the CDC Spanish-language tri-fold brochure titled Screen for Life and an I-FOBT card. The participant will be instructed to review the materials in clinic and complete the I-FOBT stool sampling at home. This brochure describes CRC, risk factors, symptoms, screening tests, benefits of screening, and insurance coverage.
  Interventions: Other: Immunochemical Fecal Occult Blood Test (I-FOBT) Kit; Behavioral: Standard Intervention

INTERVENTIONS:
Other: Immunochemical Fecal Occult Blood Test (I-FOBT) Kit — Both intervention groups will receive an I-FOBT kit (by study coordinator) with verbal and written instructions in Spanish on how to complete the stool sampling at home within 1 week, and mail the completed kit in the pre-addressed, postage paid mailer. Patients with abnormal results will receive a call explaining the meaning of an abnormal I-FOBT and encouraging them to take specific next steps.
Behavioral: LATINOS CARES Toolkit — DVD + photonovella booklet), about colorectal cancer screening (CRCS) targeted for a Latino medically underserved population.
  Arms: LATINOS CARES Toolkit
Behavioral: Standard Intervention — Standard intervention (CDC brochure) on colorectal cancer screening in community health clinics.
  Arms: Standard Intervention (SI)

SUMMARY:
The purpose of this study is to conduct 4 focus groups and recruit for 12 participants per focus group to explore community members' views about colorectal cancer screening (CRCS) processes and perceived benefits and impediments, what information they believe should be communicated, communication preferences (style, tone) and perceptions of screenings.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, age 50-75 years
* Self-identify as Hispanic/Latino
* Able to understand, read, and speak Spanish
* Prefer to receive health information in Spanish
* Previously screened or not screened

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2014-04-28 (Actual); Primary Completion 2016-07-14 (Actual); Study Completion 2022-10-26 (Actual)

PRIMARY OUTCOMES:
Rate of Feedback from Community Advisory Board | Up to 4 months
  Successful collection of feedback to complete production of Spanish-language LATINOS CARES Intervention.
  This aim involves no statistical analysis except the summary statistics for the participants. To adapt (transcreate) and produce an educational intervention entitled LATINOS CARES (DVD + photonovella booklet), about colorectal cancer screening (CRCS) targeted for a Latino medically underserved population. BENCHMARK: Production of Spanish-language LATINOS CARES intervention that is easy-to understand, salient, and culturally suitable.

SECONDARY OUTCOMES:
Rate of Receipt of I-FOBT from Participants | Up to 4 months
  BENCHMARK: Receipt of Immunochemical Fecal Occult Blood Test (I-FOBT home kit).
Rate of Receipt of Assessments from Participants | Up to 4 months
  BENCHMARK: Receipt of Assessments.

CONTACTS AND LOCATIONS:
Overall Officials: Clement Gwede, Ph.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States

REFERENCES:
- [Derived] Chavarria EA, Christy SM, Feng H, Miao H, Abdulla R, Gutierrez L, Lopez D, Sanchez J, Gwede CK, Meade CD. Online Health Information Seeking and eHealth Literacy Among Spanish Language-Dominant Latino Adults Receiving Care in a Community Clinic: Secondary Analysis of Pilot Randomized Controlled Trial Data. JMIR Form Res. 2022 Oct 13;6(10):e37687. doi: 10.2196/37687. PMID 35238785
- [Derived] Christy SM, Cousin LA, Sutton SK, Chavarria EA, Abdulla R, Gutierrez L, Sanchez J, Lopez D, Gwede CK, Meade CD. Characterizing Health Literacy Among Spanish Language-Preferring Latinos Ages 50-75. Nurs Res. 2021 Set/Oct 01;70(5):344-353. doi: 10.1097/NNR.0000000000000519. PMID 33990120
- See also: Moffitt Cancer Center Clinical Trials website — https://moffitt.org/